CLINICAL TRIAL: NCT05148312
Title: A Randomized, Open Label, Single-center, Single-dose, Four-period Crossover Clinical Trial to Assess the PK Profile and Safety of Budesonide Inhalation Solution AQ001S Compared to Budesonide Inhalation Suspension in Healthy Volunteers
Brief Title: Single-dose AQ001S PK Study in Healthy Volunteers
Acronym: BORA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aquilon Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BORA Study
Record Dates: First submitted 2021-11-02; First posted 2021-12-08 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2021-11

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: The study drug will be administered by nebulization. The subjects will adhere to the following therapeutic scheme at each treatment period of 3 days, for 4 treatment periods:
  * One single dose of study medication on the first day of the treatment period, followed by
  * Minimum washout period of 3 days, i.e. minimum 72 hours between two drug administrations
  The pharmacokinetics profile of budesonide in plasma, will be evaluated through pharmacokinetics parameters, calculated for each single dose, and based on 17 timepoints from 0 to 24h.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AQ001S 0.125 mg/2mL single-dose (Experimental): AQ001S 0.125 mg/2 ml (budesonide 0.125 mg/2 ml inhalation solution) single-dose administered by nebulization.
  Interventions: Drug: Budesonide Inhalant Product
- AQ001S 0.250 mg/2mL single-dose (Experimental): AQ001S 0.250 mg/2 ml (budesonide 0.250 mg/2 ml inhalation solution) single-dose administered by nebulization.
  Interventions: Drug: Budesonide Inhalant Product
- AQ001S 0.500 mg/2mL single-dose (Experimental): AQ001S 0.500 mg/2 ml (budesonide 0.500 mg/2 ml inhalation solution) single-dose administered by nebulization.
  Interventions: Drug: Budesonide Inhalant Product
- Budesonide inhalation suspension 1.0 mg/2 ml single-dose (Active Comparator): Pulmicort Respules® 1.0 mg/2 ml is a budesonide inhalation suspension administered by nebulization.
  Interventions: Drug: Budesonide Inhalant Product

INTERVENTIONS:
Drug: Budesonide Inhalant Product — Single-dose of budesonide solution administered by nebulization.
  Other Names: Budesonide solution administered by nebulization

SUMMARY:
This is a randomized, open label, single-center, single-dose, four-period crossover clinical study to assess the pharmacokinetic profile and safety of a budesonide inhalation solution (AQ001S) compared to a budesonide inhalation suspension (comparator) in healthy volunteers.

DETAILED DESCRIPTION:
This is a randomized, open label, single-center, single-dose, four-period crossover clinical study to assess the pharmacokinetic profile and safety of a budesonide inhalation solution (AQ001S) compared to a budesonide inhalation suspension (comparator) in healthy volunteers. Three (3) different AQ001S concentrations (i.e. 0.125 mg/2 mL, 0.250 mg/2mL and 0.500 mg/2 mL) will be compared to budesonide inhalation suspension 1.0 mg/2 ml.

Twenty (20) male and female healthy volunteers, from 18 to 60 years old, must complete the study. The study drug will be administered by nebulization.

The primary PK objective is to characterize the pharmacokinetic (PK) profile of AQ001S inhalation solution.

The primary safety objective is to assess the safety of AQ001S inhalation solution.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have given written informed consent.
2. Healthy volunteers of both genders, aged ≥ 18 and ≤ 60 years.
3. Subjects with body weight > 45 kg and Body Mass Index ≥ 18.5 and ≤ 24.9kg/m2.
4. Healthy volunteers are declared healthy based on medical history, physical examination, electrocardiogram, pulmonary function test (Forced Expiratory Volume in 1 second ≥ 80% of the predicted normal value and Forced Expiratory Volume in 1 second/ Forced Vital Capacity ≥ 70%).
5. Clinical laboratory values within the laboratory stated normal range; if not within this range, they must be without any clinical significance according to the Investigator.
6. Subjects who never smoked.
7. Women of childbearing potential (WOCBP) may be enrolled if they practice a method of birth control with a reliability of at least 90% and agree to continue doing so throughout the treatment period (e.g. condom, intrauterine device or hormonal contraception).
8. Any female subject with childbearing potential has a negative pregnancy test at Screening visit and prior to dosing at each treatment period.
9. Reliable subjects who are willing to be available for the duration of the clinical study and willing to comply with clinical study procedures.
10. Subjects who have the ability to understand the requirements of the clinical study.

Exclusion Criteria:

1. Any clinically important abnormality identified at the screening medical assessment (physical examination/medical history) or clinically relevant laboratory abnormalities.
2. Clinically significant history or presence of pulmonary malformations, chronic bronchitis, asthma, emphysema, cystic fibrosis or any other pulmonary disease
3. History or presence of pulmonary tuberculosis.
4. Viral or bacterial upper or lower respiratory tract infection, or sinus or middle ear infection, within 4 weeks prior to the screening visit.
5. Untreated oral candidiasis.
6. History or presence of prolonged QTc interval (> 450 ms), or any other clinically significant electrocardiogram abnormalities as judged by the Investigator based on 12-lead electrocardiogram recordings at Screening Visit.
7. History or presence of malignancy of any system organ class (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years prior to Screening Visit, regardless of whether there is no evidence of local recurrence or metastases.
8. Eye disorders, especially glaucoma, or a family history of glaucoma.
9. History of alcohol or drug abuse.
10. Inability to abstain from alcohol consumption for the duration of study period.
11. Immunosuppressive treatment, including topical and systemic corticosteroids (e.g., oral, parenteral, ocular, nasal or inhaled), within 4 weeks before Screening Visit.
12. Use of prescription or non-prescription drugs, except for simple analgesics (e.g. paracetamol) and hormonal contraception for women, including vitamins, herbal and dietary supplements (including St John's Wort [Hypericum]) within 7 days (or 2 weeks if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before the Screening Visit.
13. Pregnant or breastfeeding female subjects.
14. History of hypersensitivity or existing contraindication to budesonide or any other study medication ingredients.
15. Blood or plasma donation within 4 weeks prior to Screening Visit.
16. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the clinical study.
17. History or presence of any other clinically relevant disease of any major system organ class (e.g. cardiovascular, pulmonary, renal, hepatic, gastrointestinal, reproductive, endocrinological including any type of Diabetes mellitus, neurological, psychiatric or orthopedic disease) as judged by the Investigator.
18. COVID-19, Hepatitis B and C and HIV positive tests
19. Any COVID-19 vaccine within 2 weeks prior to the first dose of study drugs, and during the entire study participation including 2 weeks after the last dose of study drug.
20. Subjects who participated in an investigational study within the 12 weeks prior to the start of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacokinetics (Cmax) of budesonide through analysis of blood samples | Day 1 (predose) and at 2', 5', 10', 15', 20', 30', 45', 60', 90', 120', 180', 240', 360', 10h, 18h and 24h postdose
  Blood samples will be collected from each subject using an indwelling intravenous catheter.
  In total 17 blood samples for PK assessments over 24 hours will be collected.
Assessment of pharmacokinetics (Tmax) of budesonide through analysis of blood samples | Day 1 (predose) and at 2', 5', 10', 15', 20', 30', 45', 60', 90', 120', 180', 240', 360', 10h, 18h and 24h postdose
  Blood samples will be collected from each subject using an indwelling intravenous catheter.
  In total 17 blood samples for PK assessments over 24 hours will be collected.
Assessment of pharmacokinetics (AUC) of budesonide through analysis of blood samples | Day 1 (predose) and at 2', 5', 10', 15', 20', 30', 45', 60', 90', 120', 180', 240', 360', 10h, 18h and 24h postdose
  Blood samples will be collected from each subject using an indwelling intravenous catheter.
  In total 17 blood samples for PK assessments over 24 hours will be collected.
Assessment of the safety through to incidence of Adverse Events of AQ001S inhalation solution | From baseline up to 17 days after first study drug intake
  Incidence of treatment-related adverse events (AE), including acute bronchospasm
Assessment of the general tolerability through to vital signs (blood pressure: systolic and diastolic blood pressure) of AQ001S inhalation solution | From baseline up to 17 days after first study drug intake
  Vital signs assessment through blood pressure (systolic and diastolic blood pressure)
Assessment of the general tolerability through to vital signs (pulse rate) of AQ001S inhalation solution | From baseline up to 17 days after first study drug intake
  Vital signs assessment through pulse rate
Assessment of the general tolerability through to vital signs (respiratory rate) of AQ001S inhalation solution | From baseline up to 17 days after first study drug intake
  Vital signs assessment through respiratory rate
Assessment of the general tolerability through to ECG (PR interval duration) | From baseline up to 17 days after first study drug intake
  ECG assessment through to PR interval duration
Assessment of the general tolerability through to ECG (heart rhythm) of AQ001S inhalation solution | From baseline up to 17 days after first study drug intake
  ECG assessment through to heart rhythm
Assessment of the general tolerability through to ECG (QRS interval duration) of AQ001S inhalation solution | From baseline up to 17 days after first study drug intake
  ECG assessment through to QRS interval duration
Assessment of the general tolerability through to ECG (Corrected QT interval (QTc)) of AQ001S inhalation solution | From baseline up to 17 days after first study drug intake
  ECG assessment through to Corrected QT interval
Assessment of the general tolerability through to ECG (QT interval duration) of AQ001S inhalation solution | From baseline up to 17 days after first study drug intake
  ECG assessment through to QT interval duration
Assessment of the general tolerability through to physical examination | From baseline up to 17 days after first study drug intake
  General tolerability through the rate of patients with observed abnormalities in the following organic systems: general appearance, head and neck (incl. oropharyngeal examination), skin, respiratory system, cardiovascular system, abdomen, urogenital system, nervous system, ear, eyes and nose, musculoskeletal system
Assessment of the local tolerability through to increased bronchial irritability of AQ001S inhalation solution | From baseline up to 17 days after first study drug intake
  Incidence of Increased bronchial irritability
Assessment of the local tolerability through to paradoxical bronchospasm of AQ001S inhalation solution | From baseline up to 17 days after first study drug intake
  Incidence of paradoxical bronchospasm
Assessment of the local tolerability through to oropharyngeal examination ((e.g. vocal cord myopathy, fungal infection) of AQ001S inhalation solution | From baseline up to 17 days after first study drug intake
  Incidence of oropharyngeal examination ((e.g. vocal cord myopathy, fungal infection)

CONTACTS AND LOCATIONS:
Overall Officials: Dobrin Svinarov, MD, Principal Investigator — MC Comac Medical Ltd.
Locations (1):
- MC Comac Medical Ltd., Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, CSR
Time Frame: Beginning 6 months and ending 5 years following article publication.
Access Criteria: To Investigators whose proposed use of the data has been approved by sponsor.